CLINICAL TRIAL: NCT05534412
Title: A Practice-Based Intervention to Improve Care for a Diverse Population of Women with Urinary Incontinence
Acronym: OPTIMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Cedars-Sinai Medical Center (Other); University of California, Los Angeles (Other); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); RAND (Other)
Responsible Party: Principal Investigator, Jennifer Anger, Professor of Urology, Vice Chair of Research, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 802004
Record Dates: First submitted 2022-08-01; First posted 2022-09-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Urinary Incontinence
Keywords: Practice-based intervention; Patient-centered outcomes research; Disparities; Quality of care indicators; Primary care; Urinary incontinence; Stress incontinence; Urge incontinence; Mixed incontinence; Overactive bladder
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Urinary Incontinence, Urge; Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Four Southern California medical groups will participate in a cluster randomized controlled trial in which 60 offices (15 per site) will be randomized to undergo a practice-based incontinence intervention or control for 6 months. After the study trial, the control offices will then undergo the intervention as part of a "validation phase" of the study.
Who Masked: Participant
Masking Description: Patients will be aware that their primary care physician is participating in the study. However, they will not be informed of which arm the physician belongs to. Primary care physicians will be aware of which arm their office was assigned to based on whether or not they receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Practice-Based Intervention (Experimental): The intervention will include physician education, electronic decision support, implementation of an electronic referral system, and patient education/co-management by an advance practice provider.
  Interventions: Other: Academic Detailing; Other: Electronic Clinical Decision Support; Other: APP Co-management; Other: Electronic Referral
- Control (No Intervention): Offices in this group will not receive the four-pronged intervention. However, after the study trial, there will be a "validation phase" in which the initial control group will then receive the intervention. This cross-over deign will then allow all 60 offices to receive the intervention. Data from the cross-over intervention group will be analyzed as a separate cohort to confirm improvements in patient care and outcomes as measured in the intervention group under the study trial can be duplicated.

INTERVENTIONS:
Other: Academic Detailing — 1. Provider Assessment. Physicians and advance practice providers will complete questionnaires before the intervention that assess their knowledge about the treatment for UI in women.
  2. Mealtime Lecture. A group meeting will take place for the physicians in the intervention groups. All aspects of incontinence care will be addressed-including elements of the history and physical examination, initiation of conservative treatment, as well as when to refer for second-line therapies performed by specialists-utilizing the the principles of Academic Detailing.
  3. Monthly individual feedback. Physicians and their clinical champion specialist will meet for individual coaching one month after the mealtime lecture to discuss and review the physician's previous performance as measured by the baseline chart abstraction. Physicians will have monthly check-ins with their clinical champion via a combination of quarterly synchronous Zooms and monthly asynchronous emails.
  Arms: Practice-Based Intervention
Other: Electronic Clinical Decision Support — Intervention physicians will have access to electronic clinical decision support consisting of note templates, order sets, interruptive alerts, and a notification of patients who screen positive for UI.
  Arms: Practice-Based Intervention
Other: APP Co-management — To reduce additional burden of care on the PCPs, the investigators will incorporate Advanced Practices Providers into the patient education and self-management portion of care. The APPs will be trained together with the intervention physicians, but they will also undergo additional standardized training on patient education, UI knowledge, providing instruction on Kegel exercises, shared decision making, and self management.
  Patients will then be scheduled for a UI education and self-management session with the APP by telemedicine (video visit or telephone visit) within one month of their initial visit. For patients in need of an annual pelvic examination, and if the patient's PCP prefers to have the APP conduct the pelvic exam, a separate visit will be scheduled with the APP. A followup televisit will then be scheduled within three months of the initial APP visit, in order to assess the outcome of non-surgical treatment and determine if a specialist referral is indicated.
  Arms: Practice-Based Intervention
Other: Electronic Referral — In implementing the electronic consultation system in the private sector, the investigators will model the Expected Practice developed by the Los Angeles County Specialty-Primary Care Work Group. This eConsult system utilizes a "kickback" mechanism by which a specialist, who reviews the referral, can return it if it has not met certain baseline criteria (e.g. for a woman with OAB/urinary urgency: document negative UA, scheduled voids, titrate fluids to thirst, Kegels, antimuscarinics, optimize diuretic control, adjust any diuretics).
  Arms: Practice-Based Intervention

SUMMARY:
The main goal of this clinical trial is to improve the care for urinary incontinence (UI) provided to adult women by primary care providers. The main questions it aims to answer are:

* Can a practice-based intervention involving primary care providers lead to improved quality of incontinence care?
* Will this intervention reduce the utilization of specialist care for urinary incontinence?
* What effect will this intervention have on patient outcomes, including disease-specific outcomes, symptom severity, quality of life, and patient knowledge?
* Does our intervention reduce disparities in care?

Provider participants will be randomized at the office level to either an intervention group or a delayed intervention (control) group. The intervention group will receive an intervention consisting of academic detailing, clinical decision support tools, electronic referral, and the ability to refer to an advanced practice provider for co-management. The delayed intervention group will provide usual care until the crossover phase of the study, at which point they will receive the same intervention as the intervention group.

Patient participants will bring up urinary incontinence with their primary care provider and complete three electronic surveys.

Researchers will compare the intervention group to the delayed intervention (control) group to see if the intervention results in increased adherence to evidence-based quality indicators.

DETAILED DESCRIPTION:
The burden of urinary incontinence (UI) on American women is immense in human and financial terms, and continues to rise with the growing population of older adults. The goal of this proposal is to improve the care for UI provided to women and, in doing so, decrease the utilization of specialty care while improving patient outcomes. Specific Aim 1 seeks to improve the quality of incontinence care provided to an ethnically diverse population of women through a controlled practice-based intervention involving primary care providers. The intervention involves the implementation of PCOR measures. Four Southern California medical groups will participate in a cluster randomized controlled trial in which 60 offices (15 per site) will be randomized to undergo a practice-based incontinence intervention led by a "clinical champion dyad" comprised of a primary care provider and urologist/urogynecologist, both of whom are members of that specific medical group. The intervention will include physician education, individual performance feedback, electronic decision support, patient education using dedicated advanced practice providers (APPs), and the implementation of an electronic referral service. The quality of patient care, as evidenced by compliance with primary care UI quality indicators the investigators developed and pilot-tested, will be measured across the two randomized arms after implementation of the intervention. Compliance with these quality indicators will be the key means to implement PCOR evidence, while, at the same time, measure quality. In Specific Aim 2, utilization of specialists will be compared before and after the intervention. The investigators hypothesize that improved care at the level of the primary care physician will reduce the number of specialty referrals. Specific Aim 3 will seek to measure the effect of the intervention on patient outcomes. Under the hypothesis that a practice-based intervention will improve disease-specific outcomes, symptom severity, quality of life, and patient knowledge will be measured at baseline using validated questionnaires. After implementation of the intervention, these questionnaires will be given a second time six months later and outcomes will be compared between control and intervention groups. The investigators expect that this intervention will also reduce disparities in care for underrepresented minorities.

ELIGIBILITY:
Inclusion Criteria of Primary Care Physicians:

* Primary care physician belonging to a recruited office among one of four participating sites: Cedars-Sinai, Harbor-UCLA, UCLA, UCSD

Inclusion Criteria of Patients

* Age >18 y/o
* English or Spanish fluency
* Female
* Answers "yes" to incontinence screening tool and agrees to participate

Exclusion Criteria of Primary Care Physicians:

* Non-primary care specialty
* Does not belong to one of the participating offices

Exclusion Criteria of Patients

* Age <18 y/o
* Answers "no" to incontinence screening tool and/or does not agree to participate
* Patient seen by a urinary incontinence specialist (urologist/urogynecologist) for urinary incontinence in the past two years
* Primary care provider (who reviews a list of patients that screen positive) deems patient ineligible due to pregnant, severe memory impairment, or psychiatric history preventing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Adherence to evidence-based quality-of-care indicators | Baseline, 3 months, 6 months
  Adherence to the QIs for patients who screen positive for UI will be compared across the two randomized arms at baseline and again at 3 and 6 months after intervention implementation.

SECONDARY OUTCOMES:
Referral rates to a specialist | Baseline, 6 months
  The number of referrals to a specialist over the intervention period (urologist or gynecologist) will be quantified and compared between intervention and control groups.
  For patients screened as positive for new or worsening UI at their primary care physician office from Specific Aim 1, the investigators will record if and when the patient was referred to a specialist for treatment. Dates of each level of care provided will be incorporated into each chart abstraction so that the timing can be calculated. Investigators will also record the baseline rate of specialty referrals for each office during the baseline chart review.
ICIQ-SF | Baseline, 3 months, 6 months
  Four-item questionnaire that evaluates frequency, severity and impact on quality of life of UI.
UDI-6 | Baseline, 3 months, 6 months
  Six-item questionnaire that measures quality of life and symptom distress for UI in women.
PGI-I | 3 months, 6 months
  Global index (transition scale) that measures symptom improvement.
PFAKS | Baseline, 6 months
  Thirty-one-item questionnaire assessing patient knowledge in three domains: POP (11 items), SUI (10 items) and OAB (10 items) with questions on condition pathophysiology, management, and quality of life.
SDM-Q-9 | 6 months
  Nine-item questionnaire that measures the extent to which patients are involved in the process of decision-making.
Net Promoter Score | 3 months, 6 months
  Single-item questionnaire to evaluate the patient's willingness to refer their provider to a friend
IIQ-7 | Baseline, 3 months, 6 months
  Seven-item questionnaire to assess quality-of-life impact of UI

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California, San Diego, La Jolla, California
  - Cedars-Sinai, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Harbor-UCLA Medical Center, Torrance, California

IPD SHARING:
Plan to Share IPD: Yes
Available by request.

REFERENCES:
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Am J Obstet Gynecol. 2002 Jul;187(1):116-26. doi: 10.1067/mob.2002.125704. No abstract available. PMID 12114899
- [Background] Markland AD, Richter HE, Fwu CW, Eggers P, Kusek JW. Prevalence and trends of urinary incontinence in adults in the United States, 2001 to 2008. J Urol. 2011 Aug;186(2):589-93. doi: 10.1016/j.juro.2011.03.114. PMID 21684555
- [Background] Dieter AA, Wilkins MF, Wu JM. Epidemiological trends and future care needs for pelvic floor disorders. Curr Opin Obstet Gynecol. 2015 Oct;27(5):380-4. doi: 10.1097/GCO.0000000000000200. PMID 26308198
- [Background] Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6. doi: 10.1016/S0029-7844(97)00058-6. PMID 9083302
- [Background] L.A. WL. Race Ethnicity Pie Chart. Available from: https://www.welikela.com/wpcontent/uploads/2020/05/race-ethnicity-pie-chart.png.
- [Background] Anger JT, Saigal CS, Litwin MS; Urologic Diseases of America Project. The prevalence of urinary incontinence among community dwelling adult women: results from the National Health and Nutrition Examination Survey. J Urol. 2006 Feb;175(2):601-4. doi: 10.1016/S0022-5347(05)00242-9. PMID 16407004
- [Background] Wu JM, Hundley AF, Fulton RG, Myers ER. Forecasting the prevalence of pelvic floor disorders in U.S. Women: 2010 to 2050. Obstet Gynecol. 2009 Dec;114(6):1278-1283. doi: 10.1097/AOG.0b013e3181c2ce96. PMID 19935030
- [Background] Mesens T, Aich A, Bhal PS. Late erosions of mid-urethral tapes for stress urinary incontinence--need for long-term follow-up? Int Urogynecol J Pelvic Floor Dysfunct. 2007 Sep;18(9):1113-4. doi: 10.1007/s00192-007-0301-4. Epub 2007 Mar 9. PMID 17347793
- [Background] Schnelle JF, Smith RL. Quality indicators for the management of urinary incontinence in vulnerable community-dwelling elders. Ann Intern Med. 2001 Oct 16;135(8 Pt 2):752-8. doi: 10.7326/0003-4819-135-8_part_2-200110161-00015. No abstract available. PMID 11601959
- [Background] Gnanadesigan N, Saliba D, Roth CP, Solomon DH, Chang JT, Schnelle J, Smith R, Shekelle PG, Wenger NS. The quality of care provided to vulnerable older community-based patients with urinary incontinence. J Am Med Dir Assoc. 2004 May-Jun;5(3):141-6. doi: 10.1097/01.JAM.0000123026.47700.1A. PMID 15115573
- [Background] Anger JT, Alas A, Litwin MS, Chu SD, Bresee C, Roth CP, Rashid R, Shekelle P, Wenger NS. The Quality of Care Provided to Women with Urinary Incontinence in 2 Clinical Settings. J Urol. 2016 Oct;196(4):1196-200. doi: 10.1016/j.juro.2016.05.005. Epub 2016 May 7. PMID 27164512
- [Background] Shi L. The impact of primary care: a focused review. Scientifica (Cairo). 2012;2012:432892. doi: 10.6064/2012/432892. Epub 2012 Dec 31. PMID 24278694
- [Background] Daneshgari F, Imrey PB, Risendal B, Dwyer A, Barber MD, Byers T. Differences in urinary incontinence between Hispanic and non-Hispanic white women: a population-based study. BJU Int. 2008 Mar;101(5):575-9. doi: 10.1111/j.1464-410X.2007.07333.x. Epub 2008 Jan 8. PMID 18190644
- [Background] Anger JT, Rodriguez LV, Wang Q, Chen E, Pashos CL, Litwin MS. Racial disparities in the surgical management of stress incontinence among female Medicare beneficiaries. J Urol. 2007 May;177(5):1846-50. doi: 10.1016/j.juro.2007.01.035. PMID 17437833
- [Background] Alas AN, Dunivan GC, Wieslander CK, Sevilla C, Barrera B, Rashid R, Maliski S, Eilber K, Rogers RG, Anger JT. Health Care Disparities Among English-Speaking and Spanish-Speaking Women With Pelvic Organ Prolapse at Public and Private Hospitals: What Are the Barriers? Female Pelvic Med Reconstr Surg. 2016 Nov/Dec;22(6):460-466. doi: 10.1097/SPV.0000000000000315. PMID 27636216
- [Background] Reuben DB, Roth C, Kamberg C, Wenger NS. Restructuring primary care practices to manage geriatric syndromes: the ACOVE-2 intervention. J Am Geriatr Soc. 2003 Dec;51(12):1787-93. doi: 10.1046/j.1532-5415.2003.51565.x. PMID 14687359
- [Background] Min LC, Reuben DB, Adams J, Shekelle PG, Ganz DA, Roth CP, Wenger NS. Does better quality of care for falls and urinary incontinence result in better participant-reported outcomes? J Am Geriatr Soc. 2011 Aug;59(8):1435-43. doi: 10.1111/j.1532-5415.2011.03517.x. Epub 2011 Aug 1. PMID 21806560
- [Background] Soumerai SB, Avorn J. Principles of educational outreach ('academic detailing') to improve clinical decision making. JAMA. 1990 Jan 26;263(4):549-56. PMID 2104640
- [Background] Rugh JD, Sever N, Glass BJ, Matteson SR. Transferring evidence-based information from dental school to practitioners: a pilot "academic detailing" program involving dental students. J Dent Educ. 2011 Oct;75(10):1316-22. PMID 22012774
- [Background] O'Brien MA, Rogers S, Jamtvedt G, Oxman AD, Odgaard-Jensen J, Kristoffersen DT, Forsetlund L, Bainbridge D, Freemantle N, Davis DA, Haynes RB, Harvey EL. Educational outreach visits: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD000409. doi: 10.1002/14651858.CD000409.pub2. PMID 17943742
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness. JAMA. 2002 Oct 9;288(14):1775-9. doi: 10.1001/jama.288.14.1775. PMID 12365965
- [Background] Wagner EH. Chronic disease management: what will it take to improve care for chronic illness? Eff Clin Pract. 1998 Aug-Sep;1(1):2-4. No abstract available. PMID 10345255
- [Background] Coleman K, Austin BT, Brach C, Wagner EH. Evidence on the Chronic Care Model in the new millennium. Health Aff (Millwood). 2009 Jan-Feb;28(1):75-85. doi: 10.1377/hlthaff.28.1.75. PMID 19124857
- [Background] Anger JT, Scott VC, Kiyosaki K, Khan AA, Weinberg A, Connor SE, Roth CP, Wenger N, Shekelle P, Litwin MS. Development of quality indicators for women with urinary incontinence. Neurourol Urodyn. 2013 Nov;32(8):1058-63. doi: 10.1002/nau.22353. Epub 2013 Sep 16. PMID 24105879
- [Background] Wenger NS, Roth CP, Shekelle PG, Young RT, Solomon DH, Kamberg CJ, Chang JT, Louie R, Higashi T, MacLean CH, Adams J, Min LC, Ransohoff K, Hoffing M, Reuben DB. A practice-based intervention to improve primary care for falls, urinary incontinence, and dementia. J Am Geriatr Soc. 2009 Mar;57(3):547-55. doi: 10.1111/j.1532-5415.2008.02128.x. Epub 2009 Jan 16. PMID 19175441
- [Background] Smith AL, Nissim HA, Le TX, Khan A, Maliski SL, Litwin MS, Sarkisian CA, Raz S, Rodriguez LV, Anger JT. Misconceptions and miscommunication among aging women with overactive bladder symptoms. Urology. 2011 Jan;77(1):55-9. doi: 10.1016/j.urology.2010.07.460. Epub 2010 Oct 23. PMID 20970839
- [Background] Brook RH, Chassin MR, Fink A, Solomon DH, Kosecoff J, Park RE. A method for the detailed assessment of the appropriateness of medical technologies. Int J Technol Assess Health Care. 1986;2(1):53-63. doi: 10.1017/s0266462300002774. No abstract available. PMID 10300718
- [Background] Shekelle PG, Chassin MR, Park RE. Assessing the predictive validity of the RAND/UCLA appropriateness method criteria for performing carotid endarterectomy. Int J Technol Assess Health Care. 1998 Fall;14(4):707-27. doi: 10.1017/s0266462300012022. PMID 9885461
- [Background] Kravitz RL, Park RE, Kahan JP. Measuring the clinical consistency of panelists' appropriateness ratings: the case of coronary artery bypass surgery. Health Policy. 1997 Nov;42(2):135-43. doi: 10.1016/s0168-8510(97)00064-x. PMID 10175621
- [Background] Qaseem A, Dallas P, Forciea MA, Starkey M, Denberg TD, Shekelle P; Clinical Guidelines Committee of the American College of Physicians. Nonsurgical management of urinary incontinence in women: a clinical practice guideline from the American College of Physicians. Ann Intern Med. 2014 Sep 16;161(6):429-40. doi: 10.7326/M13-2410. PMID 25222388
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Kellogg KM, Hettinger Z, Shah M, Wears RL, Sellers CR, Squires M, Fairbanks RJ. Our current approach to root cause analysis: is it contributing to our failure to improve patient safety? BMJ Qual Saf. 2017 May;26(5):381-387. doi: 10.1136/bmjqs-2016-005991. Epub 2016 Dec 9. PMID 27940638
- [Background] Wenger NS, Roth CP, Hall WJ, Ganz DA, Snow V, Byrkit J, Dzielak E, Gullen DJ, Loepfe TR, Sahler C, Snooks Q, Beckman R, Adams J, Rosen M, Reuben DB. Practice redesign to improve care for falls and urinary incontinence: primary care intervention for older patients. Arch Intern Med. 2010 Oct 25;170(19):1765-72. doi: 10.1001/archinternmed.2010.387. PMID 20975026
- [Background] Miller DC, Murtagh DS, Suh RS, Knapp PM, Dunn RL, Montie JE. Establishment of a urological surgery quality collaborative. J Urol. 2010 Dec;184(6):2485-90. doi: 10.1016/j.juro.2010.08.015. Epub 2010 Oct 18. PMID 20961582
- [Background] Miller DC, Murtagh DS, Suh RS, Knapp PM, Schuster TG, Dunn RL, Montie JE. Regional collaboration to improve radiographic staging practices among men with early stage prostate cancer. J Urol. 2011 Sep;186(3):844-9. doi: 10.1016/j.juro.2011.04.078. Epub 2011 Jul 23. PMID 21788043
- [Background] Charmaz K. Qualitative interviewing and grounded theory analysis. In: Gubrium JF, Holstein JA, editors. Handbook of Interview Research: Context and Method. Thousand Oaks, California: Sage Publications; 2002. p.675-94.
- [Background] Lee UJ, Scott VC, Rashid R, Behniwal A, Wein AJ, Maliski SL, Anger JT. Defining and managing overactive bladder: disagreement among the experts. Urology. 2013 Feb;81(2):257-62. doi: 10.1016/j.urology.2012.09.028. PMID 23374774
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Simon SR, Majumdar SR, Prosser LA, Salem-Schatz S, Warner C, Kleinman K, Miroshnik I, Soumerai SB. Group versus individual academic detailing to improve the use of antihypertensive medications in primary care: a cluster-randomized controlled trial. Am J Med. 2005 May;118(5):521-8. doi: 10.1016/j.amjmed.2004.12.023. PMID 15866255
- [Background] Jamtvedt G, Young JM, Kristoffersen DT, O'Brien MA, Oxman AD. Audit and feedback: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD000259. doi: 10.1002/14651858.CD000259.pub2. PMID 16625533
- [Background] Shojania KG, Jennings A, Mayhew A, Ramsay CR, Eccles MP, Grimshaw J. The effects of on-screen, point of care computer reminders on processes and outcomes of care. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD001096. doi: 10.1002/14651858.CD001096.pub2. PMID 19588323
- [Background] Bates DW, Kuperman GJ, Wang S, Gandhi T, Kittler A, Volk L, Spurr C, Khorasani R, Tanasijevic M, Middleton B. Ten commandments for effective clinical decision support: making the practice of evidence-based medicine a reality. J Am Med Inform Assoc. 2003 Nov-Dec;10(6):523-30. doi: 10.1197/jamia.M1370. Epub 2003 Aug 4. PMID 12925543
- [Background] Pevnick JM, Li X, Grein J, Bell DS, Silka P. A retrospective analysis of interruptive versus non-interruptive clinical decision support for identification of patients needing contact isolation. Appl Clin Inform. 2013 Dec 4;4(4):569-82. doi: 10.4338/ACI-2013-04-RA-0021. eCollection 2013. PMID 24454583
- [Background] Lee MS, Ray KN, Mehrotra A, Giboney P, Yee HF Jr, Barnett ML. Primary Care Practitioners' Perceptions of Electronic Consult Systems: A Qualitative Analysis. JAMA Intern Med. 2018 Jun 1;178(6):782-789. doi: 10.1001/jamainternmed.2018.0738. PMID 29801079
- [Background] Barnett ML, Yee HF Jr, Mehrotra A, Giboney P. Los Angeles Safety-Net Program eConsult System Was Rapidly Adopted And Decreased Wait Times To See Specialists. Health Aff (Millwood). 2017 Mar 1;36(3):492-499. doi: 10.1377/hlthaff.2016.1283. PMID 28264951
- [Background] Reuben DB, Ganz DA, Roth CP, McCreath HE, Ramirez KD, Wenger NS. Effect of nurse practitioner comanagement on the care of geriatric conditions. J Am Geriatr Soc. 2013 Jun;61(6):857-867. doi: 10.1111/jgs.12268. PMID 23772723
- [Background] Ganz DA, Koretz BK, Bail JK, McCreath HE, Wenger NS, Roth CP, Reuben DB. Nurse practitioner comanagement for patients in an academic geriatric practice. Am J Manag Care. 2010 Dec 1;16(12):e343-55. PMID 21291291
- [Background] O'Reilly N, Nelson HD, Conry JM, Frost J, Gregory KD, Kendig SM, Phipps M, Salganicoff A, Ramos D, Zahn C, Qaseem A; Women's Preventive Services Initiative. Screening for Urinary Incontinence in Women: A Recommendation From the Women's Preventive Services Initiative. Ann Intern Med. 2018 Sep 4;169(5):320-328. doi: 10.7326/M18-0595. Epub 2018 Aug 14. PMID 30105360
- [Background] Gallis JA, Li F, Yu H, Turner EL. cvcrand and cptest: Commands for efficient design and analysis of cluster randomized trials using constrained randomization and permutation tests. Stata J. 2018 Jun 1;18(2):357-378. doi: 10.1177/1536867x1801800204. PMID 34413708
- [Background] Zwarenstein M, Treweek S, Gagnier JJ, Altman DG, Tunis S, Haynes B, Oxman AD, Moher D; CONSORT group; Pragmatic Trials in Healthcare (Practihc) group. Improving the reporting of pragmatic trials: an extension of the CONSORT statement. BMJ. 2008 Nov 11;337:a2390. doi: 10.1136/bmj.a2390. PMID 19001484
- [Background] Wenger NS, Solomon DH, Roth CP, MacLean CH, Saliba D, Kamberg CJ, Rubenstein LZ, Young RT, Sloss EM, Louie R, Adams J, Chang JT, Venus PJ, Schnelle JF, Shekelle PG. The quality of medical care provided to vulnerable community-dwelling older patients. Ann Intern Med. 2003 Nov 4;139(9):740-7. doi: 10.7326/0003-4819-139-9-200311040-00008. PMID 14597458
- [Background] McGlynn EA, Asch SM, Adams J, Keesey J, Hicks J, DeCristofaro A, Kerr EA. The quality of health care delivered to adults in the United States. N Engl J Med. 2003 Jun 26;348(26):2635-45. doi: 10.1056/NEJMsa022615. PMID 12826639
- [Background] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571
- [Background] Hanley JA, Negassa A, Edwardes MD, Forrester JE. Statistical analysis of correlated data using generalized estimating equations: an orientation. Am J Epidemiol. 2003 Feb 15;157(4):364-75. doi: 10.1093/aje/kwf215. PMID 12578807
- [Background] Min LC, Reuben DB, MacLean CH, Shekelle PG, Solomon DH, Higashi T, Chang JT, Roth CP, Kamberg CJ, Adams J, Young RT, Wenger NS. Predictors of overall quality of care provided to vulnerable older people. J Am Geriatr Soc. 2005 Oct;53(10):1705-11. doi: 10.1111/j.1532-5415.2005.53520.x. PMID 16181169
- [Background] Campbell MK, Fayers PM, Grimshaw JM. Determinants of the intracluster correlation coefficient in cluster randomized trials: the case of implementation research. Clin Trials. 2005;2(2):99-107. doi: 10.1191/1740774505cn071oa. PMID 16279131
- [Background] Ahn C, Heo, M., and Zhang, S. . Sample Size Calculations for Clustered and Longitudinal Outcomes in Clinical Research. New York: CRC Press; 2015.
- [Background] Mueller ER, Kenton K, Tarnay C, Brubaker L, Rosenman A, Smith B, Stroupe K, Bresee C, Pantuck A, Schulam P, Anger JT. Abdominal Colpopexy: Comparison of Endoscopic Surgical Strategies (ACCESS). Contemp Clin Trials. 2012 Sep;33(5):1011-8. doi: 10.1016/j.cct.2012.05.007. Epub 2012 May 27. PMID 22643040
- [Background] Miller TA. Health literacy and adherence to medical treatment in chronic and acute illness: A meta-analysis. Patient Educ Couns. 2016 Jul;99(7):1079-1086. doi: 10.1016/j.pec.2016.01.020. Epub 2016 Feb 1. PMID 26899632
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Shumaker SA, Wyman JF, Uebersax JS, McClish D, Fantl JA. Health-related quality of life measures for women with urinary incontinence: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program in Women (CPW) Research Group. Qual Life Res. 1994 Oct;3(5):291-306. doi: 10.1007/BF00451721. PMID 7841963
- [Background] Kriston L, Scholl I, Holzel L, Simon D, Loh A, Harter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. Patient Educ Couns. 2010 Jul;80(1):94-9. doi: 10.1016/j.pec.2009.09.034. Epub 2009 Oct 30. PMID 19879711
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Background] Ruiz de Vinaspre Hernandez R, Tomas Aznar C, Rubio Aranda E. [Validation of the Spanish version of the short forms of the Urogenital Distress Inventory (UDI-6) and the Incontinence Impact Questionnaire (IIQ-7) in pregnant women]. Gac Sanit. 2011 Sep-Oct;25(5):379-84. doi: 10.1016/j.gaceta.2011.05.010. Epub 2011 Aug 25. Spanish. PMID 21871693
- [Background] Hossack T, Woo H. Validation of a patient reported outcome questionnaire for assessing success of endoscopic prostatectomy. Prostate Int. 2014 Dec;2(4):182-7. doi: 10.12954/PI.14066. Epub 2014 Dec 30. PMID 25599074
- [Background] Alvarado-Villa GE, Moncayo-Rizzo JD, Gallardo-Rumbea JA. Spanish validation endorsement of SDM-Q-9, a new approach. BMC Public Health. 2019 Jan 23;19(1):106. doi: 10.1186/s12889-019-6436-7. PMID 30674297
- See also: Care ICI. The Chronic Care Model — http://www.improvingchroniccare.org/index.php?p=the_chronic_caremodel&s=2
- See also: L.A. WL. Race Ethnicity Pie Chart. — https://www.welikela.com/wp-content/uploads/2020/05/race-ethnicity-pie-chart.png
- See also: Quality AfHRa. Nonsurgical Treatments for Urinary Incontinence in Women: A Systematic Review Update — https://effectivehealthcare.ahrq.gov/products/urinary-incontinence-update/final-report-2018
- See also: Institute P-COR. Pilot Evidence Maps: Pelvic Floor Muscle Training for Urinary Incontinence. — https://www.pcori.org/research-results/2018/pilot-evidence-maps-pelvic-floor-muscle-training-urinary-incontinence
- See also: Institute P-COR. Treating Urinary Incontinence in Women without Surgery - Evidence Update for Women — https://www.pcori.org/evidence-updates/treating-urinary-incontinence-in-women-without-surgery
- See also: CFIR Research Team-Center for Clinical Management Research. Consolidated Framework for Implementation Research (CFIR) — https://cfirguide.org
- See also: Bureau USC. QuickFacts, Los Angeles County, California — https://www.census.gov/quickfacts/fact/table/losangelescountycalifornia/AGE295220#AGE295219
- See also: Institute P-COR. Using a New Survey to Learn About Women's Experiences with Hospital Care for Childbirth — https://www.pcori.org/research-results/2017/using-new-survey-learn-about-womens-experiences-hospital-care-childbirth